CLINICAL TRIAL: NCT02699489
Title: Mansoura Enhanced Recovery Open Versus Laparoscopic Donor Nephrectomy (MEnROL): A Randomized Controlled Trial
Brief Title: Enhanced Recovery Open Versus Laparoscopic Donor Nephrectomy
Acronym: MEnROL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, ahmed mansour, Lecturer in Urology, Urology and Nephrology Center, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEnROL
Record Dates: First submitted 2016-01-13; First posted 2016-03-04 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-02

CONDITIONS: Renal Transplant Donor of Left Kidney

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopic donor nephrectomy arm (Experimental): This group will undergo laparoscopic donor nephrectomy
  Interventions: Procedure: Laparoscopic donor nephrectomy
- Open donor nephrectomy arm (Active Comparator): This group will undergo open donor nephrectomy
  Interventions: Procedure: Open donor nephrectomy

INTERVENTIONS:
Procedure: Laparoscopic donor nephrectomy — Laparoscopic donor nephrectomy performed via a standard 4-port distribution. Control of the hilar vessels is performed using extra-large Hem-o-Lok clips (Weck- Covidien, Research Triangle Park, NC) and graft extraction is performed via a pre-prepared Pfannenstiel incision
  Arms: Laparoscopic donor nephrectomy arm
Procedure: Open donor nephrectomy — Open donor nephrectomy performed via a supracostal incision above the 11th rib and an extra-pleural extra-peritoneal approach was adopted
  Arms: Open donor nephrectomy arm

SUMMARY:
A phase III randomized trial conducted to compare recovery outcomes between laparoscopic and open donor nephrectomy within a specified enhanced recovery protocol

DETAILED DESCRIPTION:
The MEnROL trial is a phase III randomized controlled trial of Open versus Laparoscopic donor nephrectomy within a standardized enhanced recovery program. Eligible donors were randomized in a 1:1 ratio.

Laparoscopic procedures are performed by a single surgeon (AMM) while Open donor nephrectomies (ODN) were performed by an experienced team that included the laparoscopic surgeon. ODN were performed via a supracostal incision above the 11th rib and an extra-pleural extra-peritoneal approach was adopted. Laparoscopic donor nephrectomy (LDN) was performed via a standard 4-port distribution. Control of the hilar vessels was performed using extra-large Hem-o-Lok clips (Weck- Covidien, Research Triangle Park, NC) and graft extraction was performed via a pre-prepared Pfannenstiel incision.

Donors are enrolled in our enhanced recovery program for donor nephrectomy. The program was compliant with the Enhanced Recovery After Surgery Group (ERAS) guidelines. All donors receive epidural analgesia and are maintained on non-narcotic postoperative analgesics. Criteria for hospital discharge include ambulation, adequate pain control with oral analgesics, and sustained intake of solid food.

ELIGIBILITY:
Inclusion Criteria:

1. Donor aged 18 years or more.
2. Donors who have the ability to understand information and materials provided.
3. Donors who didn't express a preference for either open or laparoscopic surgery.
4. Donors who are fit for both open and laparoscopic intervention
5. Donors in whom evaluation revealed left kidney with single renal artery suitable for donation.
6. Donors able to give signed written informed consent.

Exclusion Criteria:

1. Donors who had a preference for either open or laparoscopic surgery.
2. Donors in whom the right kidney was chosen for donation.
3. Donors with double renal arteries in kidneys chosen for donation.
4. Donors who didn't sign consent.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 224 (Actual)
Dates: Start 2013-01; Primary Completion 2015-06 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Donor recovery as evaluated by the physical fatigue domain of the Multidimensional Fatigue Inventory 20 (MFI-20), | 6 weeks

SECONDARY OUTCOMES:
Short Form-36 (SF-36) health survey | 6 weeks
  Scores of Short Form-36 questionnaire
Length of Hospital stay | up to 2 weeks
  Length of hospital stay in days
Ischemia times | up to 1 day
  Warm and Cold ischemia times in minutes
Duration of the procedure | up to 24 hours
  Duration of the procedure in minutes
Peri-operative complications | 90 days
  Incidence of peri-operative complications in both groups
One year graft loss | 1 year
  Incidence of one year graft loss in both groups
Recipient complications | 90 days
  Incidence of recipient complications in both groups

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data are readily shared with requesting authorities